CLINICAL TRIAL: NCT00475124
Title: VIRTUE: Virtual Clinic Pacemaker Follow-up
Brief Title: Virtual Clinic Pacemaker Follow-up
Acronym: VIRTUE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Redundant in-clinic visits increased the workload in virtual follow-up group. An interim analysis showed that the study would not support the primary hypothesis
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HS036
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Sick Sinus Syndrome; Heart Block; Bradycardia
Keywords: Pacemaker follow-up; Telecardiology; Home Monitoring
MeSH Terms: conditions — Sick Sinus Syndrome; Heart Block; Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Home Monitoring ON
  Interventions: Device: Home Monitoring of pacemaker
- 2 (Active Comparator): Home Monitoring OFF
  Interventions: Device: Home Monitoring of pacemaker deactivated

INTERVENTIONS:
Device: Home Monitoring of pacemaker — Daily Home Monitoring data transmission from the implanted pacemaker to Home Monitoring service center.
  Arms: 1
Device: Home Monitoring of pacemaker deactivated — No Home Monitoring data transmission.
  Arms: 2

SUMMARY:
Patients with implanted pacemakers are currently seen by their cardiologists every 6-12 months. Shorter follow-up intervals are generally seen as excessive workload for the physician, with little benefit for the patient. Longer intervals are seen as too dangerous concerning device integrity and safety. This scheme still results in a large number of follow-up visits with little or no important changes in pacemaker therapy.

Our clinical trial investigates efficacy and safety of the Home Monitoring technology for increasing the flexibility in pacemaker follow-up. Home Monitoring technology allows automatic transmission via mobile phone links of relevant data from the implanted pacemaker to a service center. The patient's physician can access the data via a password-protected internet site. The regular Home Monitoring data analyses entirely replace clinical routine visits ("virtual clinic"). Follow-up visits are scheduled according to the results of the Home Monitoring data analyses.

The primary endpoint of the study is to compare the total workload for pacemaker patient care in the virtual clinic with that of standard follow-up scheme with regularly scheduled clinical visits.

DETAILED DESCRIPTION:
Patients with implanted pacemakers are currently seen by their cardiologists every 6-12 months. Shorter follow-up intervals are generally seen as excessive workload for the physician, with little benefit for the patient. Longer intervals are seen as too dangerous concerning device integrity and safety. This scheme still results in a large number of follow-up visits with little or no important changes in pacemaker therapy. On the other hand, in some patients there are quicker changes in their cardiac situation and the need for subsequent adaptation of pacemaker programming, which cannot be detected and properly treated with standard follow-up scheme.

Our clinical trial investigates efficacy and safety of the Home Monitoring technology for increasing the flexibility in pacemaker follow-up. Home Monitoring technology allows automatic transmission via mobile phone links of relevant data from the implanted pacemaker to a service center. The patient's physician can access the data via a password-protected internet site. The regular Home Monitoring data analyses entirely replace clinical routine visits ("virtual clinic"). Follow-up visits are scheduled according to the results of the Home Monitoring data analyses.

For the primary endpoint, the total workload for pacemaker patient care in the virtual clinic is compared to that of a standard follow-up scheme with regular clinic visits. The total workload comprises the time for data analyses, clinical examinations, and other patient contacts.

Secondary endpoints investigate adverse events rate, quality of life, and total costs, as mirrored by direct patient's expenses, and patient travel and waiting time, for visits to the pacer clinic as well as to additional cardiologist's or internal medicine doctor's services.

Standard vs. virtual follow-up. For the standard follow-up group patients, routine follow-up visits are scheduled 1 month and 12 months after pre-discharge control, and then every 12 months. A follow-up at 6 months after discharge is optional. For the virtual clinic group patients, a routine follow-up visit is scheduled 1 month after pre-discharge control. The Home Monitoring data analyses have to be performed 12 months after discharge, and then every 12 months. If a 6-month follow-up is routinely done for the standard group in the clinic, a 6-month Home Monitoring data analysis has to be done as well. Event reports have to be analysed within 24 hours during working days.

ELIGIBILITY:
Inclusion Criteria:

* Indication for implantation of dual-chamber rate-adaptive pacemaker
* Stable medical situation
* Patient informed consent

Exclusion Criteria:

* Contra-indication for implantation of dual-chamber rate-adaptive pacemaker
* Persistent atrial fibrillation
* Replacement indication
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2007-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Total work load for virtual clinic follow-up compared to standard follow-up (without Home Monitoring) | 7 years

SECONDARY OUTCOMES:
Hospitalisation; Other serious adverse events; Quality of life; Total costs of therapy. | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: David Fluck, Dr., Study Chair — St. Peter's Hospital, Chertsey, UK
Locations (6):
- United Kingdom (6):
  - Barnet & Chase Farm Hospital, Barnet
  - Basildon Hospital, Basildon
  - St. Peter's Hospital, Chertsey
  - Russels Hall Hospital, Dudley
  - North Middlesex University Hospital, London
  - Newcross Hospital, Wolverhampton